CLINICAL TRIAL: NCT05218200
Title: The Effect of Deep Breathing and Cough Exercise on Pneumonia
Brief Title: The Effect of Deep Breathing and Cough Exercise on Respiratory Parameters in Patients With Covid-19 Associated Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Özge Uçar (Other)
Collaborators: Bartin State Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Özge Uçar, Bartın University, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-FEN-A-016
Record Dates: First submitted 2022-01-31; First posted 2022-02-01 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Pneumonia; Respiratory Disease
Keywords: Covid-19; pneumonia; breathing exercise; coughing exercise
MeSH Terms: conditions — Respiration Disorders; COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental research
Who Masked: Investigator
Masking Description: The researcher collecting data does not know the characteristics of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In addition to the routine care in the hospital, the patient will be given deep breathing and coughing exercises.
  Interventions: Other: deep breathing and coughing exercises with triflo
- Control group (No Intervention): There will be no intervention other than routine nursing care practices in the hospital.

INTERVENTIONS:
Other: deep breathing and coughing exercises with triflo — patients will be given triflo. A video of the application of deep breathing and coughing exercises with triflo prepared by the researchers will be prepared. The video will be sent to the patients' phones. It will be ensured that the patients do the exercises every hour by watching the video and they will be followed.
  Arms: experimental group

SUMMARY:
Studies reveal that the Covid-19 virus can be transmitted in three ways: respiratory tract, direct contact and feces. The incubation period is estimated to be 5.2 [4.1-7.0] days for the 95% confidence interval and the virus transmission coefficient (R0) baseline growth number is 2.2 [1.4-3.9]. The main signs and symptoms described in the literature are; other atypical symptoms, particularly fever (98%), cough (76%), myalgia or fatigue (44%); sputum (28%), headache (8%), hemoptysis (5%), vomiting (5%), diarrhea (3%) and shortness of breath were detected. In addition to lymphopenia, which is detected in 63% of cases, pneumonia is also present. Widely regarded as the cornerstone of pulmonary rehabilitation, exercise training is the best way to improve muscle function in COPD and other chronic respiratory diseases. After 326 patients hospitalized in the pandemic clinical services of a public hospital were randomly divided into the experimental (n=168) and control groups (n=168), the effect of the experiment on the respiratory parameters of the experiment will be monitored without any intervention in the control group, while deep breathing and coughing exercises will be applied to the experimental group. The aim of this study is to determine the effect of deep breathing and coughing exercises on respiratory parameters in patients treated for pneumonia due to COVID-19 disease.

DETAILED DESCRIPTION:
A new virus called SARS-CoV-2 was detected on January 7, 2020, due to the investigations carried out in the city of Wuhan, Hubei province of China, in December 2019, in 27 pneumonia cases unknown cause. The World Health Organization (WHO) declared on January 30, 2020, that it is facing a virus that threatens public health, and it was reported a pandemic on March 11, 2020.

Studies show that the virus can be transmitted in three ways: respiratory tract, direct contact, and feces.

The main signs and symptoms described in the literature are; other atypical symptoms, particularly fever (98%), cough (76%), myalgia or fatigue (44%); dyspnea (55%), sputum (28%), headache (8%), hemoptysis (5%), vomiting (5%) and diarrhea (3%). In addition to lymphopenia, which was detected in 63% of cases, all patients had pneumonia. Complications included acute respiratory distress syndrome (29%), acute heart injury (12%), and secondary infections (10%). Other more striking symptoms, such as chemosensory dysfunction, have also been described. Most of the patients diagnosed with COVID-19 have at least one underlying chronic disease (such as hypertension and chronic obstructive pulmonary disease). Many of these patients have to be treated in intensive care units (ICU). It is estimated that 80% of patients will present with mild symptoms that can be followed up without hospitalization. It is foreseen that the remaining 20% may need clinical medical care, and 5% of this may need to be hospitalized in the intensive care unit. The mean time from onset of symptoms to recovery is two weeks in patients with mild symptoms, but 3-6 weeks in patients with the severe or critical disease.

The international consensus on managing patients with Covid-19-associated acute respiratory distress syndrome (ARDS) is that despite the increasing number of reports on respiratory system mechanics and ventilation management, more experimental studies are needed. Death cases due to Covid-19 are thought to be caused mainly by ARDS. Although the incidence of ARDS reported among all Covid-19 patients is 15.6-31%, it is higher than other organ damage rates. With the increase in the number of Covid-19 patients hospitalized recently, different management strategies have started to be needed by healthcare professionals to save the lives of patients with ARDS.

In the literature, research on the pathophysiology of Covid-19 is still limited. However, evidence-based laboratory findings and clinical-pathological characteristics of Covid-19 patients suggest that secretion of large amounts of mucus in the airway interferes with the ventilation and alveolar formation process, and interstitial changes are the mechanisms underlying the impairment of gas exchange. Studies have reported that the duration of ARDS development in Covid-19 patients is between 8-12 days on average after the first symptoms are seen. Corticosteroid therapy and high-flow nasal oxygen therapy are frequently used in patients who develop ARDS. ARDS is shown as the most common cause of mortality in Covid-19 patients. Widely regarded as the cornerstone of pulmonary rehabilitation, exercise training is the best way to improve muscle function in COPD and other chronic respiratory diseases. It is indicated for patients with reduced exercise tolerance, exercise dyspnea or fatigue, impaired daily living activities, and chronic respiratory disease.

In line with these data, it is thought that specific deep breathing and coughing exercises may be beneficial to reduce reversible pulmonary changes such as secretions and interstitial fluid accumulation, maximize the area of the alveolar sacs, and accelerate the secretion clearance process.

ELIGIBILITY:
Inclusion Criteria:

* be over 18
* be conscious
* to know Turkish
* Not having any sensory or perceptual disability
* Being sick with Covid-19 pneumonia
* Volunteer

Exclusion Criteria:

* be under the age of 18
* not being conscious
* Not knowing Turkish
* Presence of any sensory or perceptual disability
* Not having covid-19 pneumonia
* Receiving mechanical ventilation support
* not volunteering

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
measuring the severity of dyspnea | 1st , 5th and 10th days
  The effect of breathing and coughing exercises with triflo on dyspnea in patients with Covid-19 pneumonia using by Dispne-12 scale.

SECONDARY OUTCOMES:
respiratory parameters | 1st, 5th and 10nd days
  The effect of deep breathing and coughing exercises with triflo on respiratory parameters in patients with Covid-19 pneumonia by using blood gas analysis result.
effect on secretion | 1st, 5th and 10nd days
  The effect of deep breathing and coughing exercises with triflo on amount of secretion in patients with Covid-19 pneumonia by using secretion measuring cup

CONTACTS AND LOCATIONS:
Overall Officials: Sevim ÇELİK, Prof., Study Director — Bartin University Health Science Faculty; Elif KARAHAN, Assoc. Prof., Study Chair — Bartin University Health Science Faculty; Suna UZUN, Study Chair — Bartin State Hospital
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No